CLINICAL TRIAL: NCT00560924
Title: Preventive Effect of Treatment With Estradiol Vaginal Tablets on Recurrent Urinary Tract Infections in Post-menopausal Women (RUTI) in Post-menopausal Women With Signs of Urogenital Ageing (UGA)
Brief Title: Preventive Effect of Treatment With Estradiol Vaginal Tablets on Recurrent Urinary Tract Infections in Post-menopausal Women
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial prematurely discontinued due to slow recruitment
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAG-1458
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Menopause; Urinary Infections
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: estradiol, 25 mcg

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the preventive effect of treatment with estradiol vaginal tablets on recurrent urinary tract infections (RUTI) in post-menopausal women with signs of urogenital ageing (UGA).

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal woman with Urogenital ageing (UGA)
* Recurrent urinary tract infections defined as three or more urinary tract infections within the past twelve months

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Present UTI
* History of RUTI during fertile period of life

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-03-21 (Actual); Primary Completion 2004-03-17 (Actual); Study Completion 2004-03-17 (Actual)

PRIMARY OUTCOMES:
Time to first symptom of urinary tract infection (UTI)

SECONDARY OUTCOMES:
Number of urinary tract infection (UTI) | During the 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Malmo, Sweden

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com